CLINICAL TRIAL: NCT06864286
Title: Effectiveness and Influencing Factors of a Nationwide Multi-dimensional Health Promotion Program for Community-Dwelling Older Adults
Brief Title: Nationwide Multi-dimensional Health Promotion Program for Community-Dwelling Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202412083RINB
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Community-dwelling Older Adults
Keywords: community-dwelling older adults; health promotion; effectiveness; influencing factors
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-domain health promotion intervention (Experimental)
  Interventions: Behavioral: Move for Health

INTERVENTIONS:
Behavioral: Move for Health — This multi-domain health promotion intervention utilizes the "Community-Based Health Promotion Program for Older Adults - Healthy Exercise Class" developed by the Health Promotion Administration (Taiwan). This intervention emphasizes a "multi-dimensional health" approach, focusing on healthy aging, exercise, and cognitive interventions, supplemented by elements of oral health, nutrition, and social participation. The program aims to promote older adults' health self-management capabilities. This 12-week program meets once weekly for two hours per session. Healthy aging curriculum covers important health issues for older adults, such as fall prevention, healthy eating, oral health, vision care, dementia prevention, medication safety, and knowledge related to healthy lifestyle behaviors including home-based exercise.

SUMMARY:
Global organizations advocate for "active" and "healthy aging," emphasizing preventive health promotion. Taiwan's Long-Term Care 2.0 and the National Health Administration's "Healthy Exercise Class" exemplify this. Evaluating these programs' effectiveness is crucial, but complex due to diverse influencing factors. This study focuses on the often-overlooked role of program leaders' facilitation skills in impacting program success.

This study investigates the effectiveness of multi-domain community health promotion programs for older adults and its influencing factors. Specifically, it aims to:

1. assess the immediate benefits (objective/subjective health status, satisfaction) for participating older adults.
2. explore related factors (group leadership skills, personal factors) using Andersen's Behavioral Model.

A prospective, single-group, pre- and post-test design will be used. Participants (leaders and older adults) will be recruited from "Healthy Exercise Class" sites nationwide. Pre- and post-intervention data will be analyzed to determine program effectiveness. Multiple linear regression will identify influencing factors, including the mediating and moderating effects of leader facilitation skill confidence. The study aims to inform policy improvements for government-led older adult health promotion.

ELIGIBILITY:
Inclusion Criteria:

- I. Leaders

1. Medical personnel (legally certified medical professionals, social workers, care service providers with licenses, and graduates of gerontological service programs) and sports professionals (National Fitness Instructors, athletic trainers, full-time sports coaches at all levels of schools, physical education teachers, professional sports background personnel with valid certificates issued by the Chinese Taipei Olympic Committee, etc.)
2. Individuals who have completed the "Basic Training Course for Sport and Health Instructors for the Prevention and Delay of Disability" offered by the Health Promotion Administration, holding a certificate of completion, or those who have been trained by local government health bureaus and passed the mutual recognition by the National Health Administration.

II. Older Adults

1. Aged 65 or above.
2. Normal cognitive function (no diagnosis of cognitive impairment-related conditions, such as mild cognitive impairment, dementia, etc.).
3. Able to communicate in Mandarin or Taiwanese.
4. Able to fully participate in the research project.

Exclusion Criteria:

- I. Leaders

1. Individuals who are unable to complete the aforementioned training program qualification or lead the program in the community.

II. Older Adults

1. Individuals whose cognitive status is affected by mental or neurological disorders, medication use, including diagnoses of mental or neurodegenerative diseases , central nervous system infections, or long-term use of medications affecting the central nervous system .
2. Individuals who meet the diagnostic criteria for mild cognitive impairment or dementia.
3. Individuals with moderate to severe disability.
4. Individuals with severe mental illness or behavioral problems (e.g., severe depression, schizophrenia, bipolar disorder, etc.).
5. Individuals who, due to visual, auditory, or physical functional impairments, are unable to complete the assessments.
6. Individuals who, due to physical or psychological illnesses, are unable to participate in the multi-domain health promotion intervention.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Study of Osteoporotic Fractures (SOF) Frailty Scale at 12 Weeks | Baseline, Week 12
  Score range: 0 to 3, with higher scores indicating worse outcomes.
Change from Baseline in the Outcome Measurement of Health-Promotion Program for Community-Dwelling Elderly at 12 Weeks | Baseline, Week 12
  The measurement includes 5 subscales: cognitive function, muscle strength, activities of daily living, nutrition, and psychosocial function.The score ranges from 0 to 100% for each subscale and the total score, with higher scores indicating better health conditions.
Change from Baseline in The Satisfaction with Life Scale at 12 Weeks | Baseline, Week 12
  Score range: 5 to 35, with higher scores indicating better outcomes.
Change from Baseline in the Self-rated Health Scale at 12 Weeks | Baseline, Week 12
  Score range: 0 to 100, with higher scores indicating better outcomes.
Course Satisfaction Questionnaire | Week 12
  Score range: 1 to 5, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Change from Baseline in the Brief Symptom Rating Scale (BSRS) at 12 Weeks | Baseline, Week 12
  Score range: 0 to 20, with higher scores indicating worse outcomes.
Change from Baseline in the Number of Self-reported Chronic Conditions at 12 Weeks | Baseline, Week 12
  A higher number of chronic conditions indicates worse outcomes.
Change from Baseline in the Body Mass Index (BMI) at 12 Weeks | Baseline, Week 12
  A BMI outside the range of 18-24 indicates worse outcomes.

OTHER OUTCOMES:
Sociodemographic Questionnaire for Older Adults | Baseline
  The questionnaire includes items such as gender, age, living status, education, marital status, employment, economic status, self-reported health conditions, activities of daily living, and transportation time to community centers.
Sociodemographic Questionnaire for Community Health Service Stations and Program Leaders | Baseline
  The questionnaire includes items such as gender, age, education, occupation, role in the community, professional background and years of experience.
Change from Baseline in the Confidence in Leadership Skills for Health Promotion Groups Questionnaire at 12 Weeks | Baseline, Week 12
  The score range is 39 to 195, with higher scores indicating greater confidence.
Change from Baseline in the Health Knowledge, Awareness and Behavior Questionnaire at 12 Weeks | Baseline, Week 12
  The score range is 31 to 124, with higher scores indicating better outcomes.
Change from Baseline in the General Self-Efficacy Scale at 12 Weeks | Baseline, Week 12
  Score range: 10 to 40, with higher scores indicating better outcomes.
Change from Baseline in the Integrated Care for Older People (ICOPE) Scale at 12 Weeks | Baseline, Week 12
  There are six key intrinsic capacities in the ICOPE, covering cognitive functions, mobility, nutrition, hearing, vision, and depression status. The ICOPE scoring results are categorized into two groups: abnormal and normal.
Participants' Attendance Rate | Every week (From Week 1 to Week 12)